CLINICAL TRIAL: NCT06420063
Title: Sequential CAR-T Cell Infusion Targeting CD33 and CD123 for Refractory/Relapsed Acute Myeloid Leukaemia
Brief Title: Sequential CAR-T Cells Targeting CD33/CD123 in Patients With Acute Myelocytic Leukemia AML
Acronym: BAH244
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202495
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: AML; Acute Myeloid Leukemia; AML, Adult Recurrent; AML, Adult
Keywords: aml; cd33; cd123; CAR-T
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this clinical trial will receive a carefully designed treatment regimen. Before the infusion of CD33 and CD123 CAR-T cells, participants will undergo preconditioning chemotherapy. This chemotherapy serves to create an optimal environment for CAR-T cell therapy to effectively target and eliminate malignant B cells. Following chemotherapy, participants will receive the infusion of CD33 and CD123 CAR-T cells.
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (CD33/CD123 CAR T cells, chemotherapy) (Experimental): Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive CD33/123 CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of CD33/123 CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of CD33/CD123 CAR T cells.
  Interventions: Biological: CD123/CD33 CART

INTERVENTIONS:
Biological: CD123/CD33 CART — The intervention in this clinical trial involves a novel approach using CD22/123-Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Patients in the trial will undergo the following regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  CD33/123-Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, CD33/123-CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial CD33/123 CAR-T cell infusion without unacceptable side effects and sufficient CAR T cell availability may receive 2 or 3 additional doses.
  Other Names: EB-BH2025

SUMMARY:
This is an open, single-arm, clinical study to evaluate the efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) targeting CD33 or CD123 or both sequentially in the treatment of Acute Myelocytic Leukemia.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. Besides CD19, many other molecules such as CD22, CD30,BCMA,CD123, etc. may have the potential to develop the corresponding CAR-T cells to treat patients whose tumors express those markers. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting CD33/CD123 in patients with Acute Myelocytic Leukemia. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, disease status after treatment will also be evaluated.

The purpose of this clinical trial is to assess the feasibility, safety, and efficacy of multiple CAR T-cell therapy which combines CAR T cells against AML Cells with CAR T cells targeting CD123 or CD33 in patients with relapsed and refractory AML. The study also aims to learn more about the function of CAR T cells and their persistence in AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute myeloid leukemia who voluntarily signed informed consent and met the following criteria:
* Age older than 6 months.
* Confirmed expression of CLL-1, CD123 and/or CD33 in blast AML by immuno-histochemical staining or flow cytometry.
* Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 3 months.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
* Hgb≥80g/L.
* No cell separation contraindications.
* Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Severe illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
* Active bacterial, fungal or viral infection not controlled by adequate treatment.
* Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Pregnant or nursing women may not participate.
* Use of glucocorticoid for systemic therapy within one week prior to entering the trial.
* Patients, in the opinion of investigators, may not be able to comply with the study.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD5/CD7 chimeric antigen receptor (CAR) T cells | 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.

SECONDARY OUTCOMES:
Rate of successful manufacture and expansion of the CD33/123 chimeric antigen receptor (CAR) T cells | 10-14 days
  satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA)

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided